CLINICAL TRIAL: NCT00300482
Title: A Multicenter, Randomized, Double-Blind, Prospective Study Comparing the Safety and Efficacy of Fenofibric Acid and Rosuvastatin Calcium Combination Therapy to Fenofibric Acid and Rosuvastatin Calcium Monotherapy in Subjects With Mixed Dyslipidemia
Brief Title: Evaluate Safety and Efficacy of ABT-335 in Combination With Rosuvastatin Calcium in Subjects With Multiple Abnormal Lipid Levels in the Blood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-748
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Dyslipidemia; Coronary Heart Disease; Mixed Dyslipidemia
Keywords: Dyslipidemia; Coronary Heart Disease; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Coronary Disease | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Active Comparator): ABT-335 + 10 mg rosuvastatin
  Interventions: Drug: ABT-335; Drug: Rosuvastatin Calcium
- B (Active Comparator): ABT-335 + 20 mg rosuvastatin
  Interventions: Drug: ABT-335; Drug: Rosuvastatin Calcium
- C (Placebo Comparator): ABT-335 monotherapy
  Interventions: Drug: ABT-335; Drug: Placebo
- D (Placebo Comparator): 10 mg rosuvastatin monotherapy
  Interventions: Drug: Rosuvastatin Calcium; Drug: Placebo
- E (Placebo Comparator): 20 mg rosuvastatin monotherapy
  Interventions: Drug: Rosuvastatin Calcium; Drug: Placebo
- F (Placebo Comparator): 40 mg rosuvastatin monotherapy
  Interventions: Drug: Rosuvastatin Calcium; Drug: Placebo

INTERVENTIONS:
Drug: ABT-335 — 135 mg, daily, 12 weeks
  Arms: A; B; C
Drug: Rosuvastatin Calcium — Daily, 12 weeks, see Arm Description for dosage information
  Other Names: Rosuvastatin
  Arms: A; B; D; E; F
Drug: Placebo — Daily, 12 weeks, see Arm Description for information regarding placebo type
  Arms: C; D; E; F

SUMMARY:
The purpose of this study is to compare the safety and efficacy of fenofibric acid (ABT-335) + rosuvastatin calcium combination therapy with ABT-335 and rosuvastatin calcium monotherapy in subjects with multiple abnormal lipid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mixed dyslipidemia

Exclusion Criteria:

* Subjects with unstable medical conditions or medical conditions considered inappropriate in a clinical trial.
* Patients who are taking certain medications or unstable dose of specific medications.
* Women who are pregnant or plan on becoming pregnant or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1445 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Kelly, MD, Principal Investigator — Abbott
Locations (1):
- Global Medical Information, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Ferdinand KC, Davidson MH, Kelly MT, Setze CM. One-year efficacy and safety of rosuvastatin + fenofibric acid combination therapy in patients with mixed dyslipidemia: evaluation of dose response. Am J Cardiovasc Drugs. 2012 Apr 1;12(2):117-25. doi: 10.2165/11597940-000000000-00000. PMID 22263674
- [Derived] Rosenson RS, Carlson DM, Kelly MT, Setze CM, Hirshberg B, Stolzenbach JC, Williams LA. Achievement of lipid targets with the combination of rosuvastatin and fenofibric Acid in patients with type 2 diabetes mellitus. Cardiovasc Drugs Ther. 2011 Feb;25(1):47-57. doi: 10.1007/s10557-010-6273-5. PMID 21174145
- [Derived] Bays HE, Roth EM, McKenney JM, Kelly MT, Thakker KM, Setze CM, Obermeyer K, Sleep DJ. The effects of fenofibric acid alone and with statins on the prevalence of metabolic syndrome and its diagnostic components in patients with mixed dyslipidemia. Diabetes Care. 2010 Sep;33(9):2113-6. doi: 10.2337/dc10-0357. Epub 2010 Jun 23. PMID 20573750
- [Derived] Jones PH, Cusi K, Davidson MH, Kelly MT, Setze CM, Thakker K, Sleep DJ, Stolzenbach JC. Efficacy and safety of fenofibric acid co-administered with low- or moderate-dose statin in patients with mixed dyslipidemia and type 2 diabetes mellitus: results of a pooled subgroup analysis from three randomized, controlled, double-blind trials. Am J Cardiovasc Drugs. 2010;10(2):73-84. doi: 10.2165/10061630-000000000-00000. PMID 20136164
- [Derived] Jones PH, Davidson MH, Kashyap ML, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Efficacy and safety of ABT-335 (fenofibric acid) in combination with rosuvastatin in patients with mixed dyslipidemia: a phase 3 study. Atherosclerosis. 2009 May;204(1):208-15. doi: 10.1016/j.atherosclerosis.2008.09.027. Epub 2008 Oct 5. PMID 18996523
- [Derived] Jones PH, Bays HE, Davidson MH, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Evaluation of a new formulation of fenofibric acid, ABT-335, co-administered with statins : study design and rationale of a phase III clinical programme. Clin Drug Investig. 2008;28(10):625-34. doi: 10.2165/00044011-200828100-00003. PMID 18783301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six subjects were randomized but not treated: 1 was lost to follow-up, 1 was randomized but deemed ineligible, 1 was withdrawn at the investigator's discretion, and 3 withdrew consent.
Groups:
- ABT-335 + 10 mg Rosuvastatin: ABT-335 + 10 mg rosuvastatin combination therapy once daily
- ABT-335 + 20 mg Rosuvastatin: ABT-335 + 20 mg rosuvastatin combination therapy once daily
- ABT-335: ABT-335 monotherapy once daily
- 10 mg Rosuvastatin: 10 mg rosuvastatin monotherapy once daily
- 20 mg Rosuvastatin: 20 mg rosuvastatin monotherapy once daily
- 40 mg Rosuvastatin: 40 mg rosuvastatin monotherapy once daily
Period: Overall Study
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Started | 261 (For all arms, "started" means treated.) | 261 | 259 | 261 | 266 | 131
Completed | 220 | 220 | 208 | 237 | 243 | 115
Not Completed | 41 | 41 | 51 | 24 | 23 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin | Total
Number analyzed (Participants) | 261 | 261 | 259 | 261 | 266 | 131 | 1439
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 206 | 209 | 209 | 222 | 217 | 103 | 1166
  >=65 years | 55 | 52 | 50 | 39 | 49 | 28 | 273
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 131 | 152 | 130 | 124 | 65 | 750
  Male | 113 | 130 | 107 | 131 | 142 | 66 | 689
Region of Enrollment [Number; unit: participants]
  North America | 261 | 261 | 259 | 261 | 266 | 131 | 1439

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Triglycerides From Baseline to Final Visit
Description: [(Week 12 triglycerides minus baseline triglycerides)/baseline triglycerides] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline triglyceride value and at least 1 postbaseline triglyceride value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 252 | 249 | 242 | 252 | 255 | 127
percent change | -47.1 (1.81) | -42.9 (1.82) | -32.6 (1.84) | -24.4 (1.81) | -25.6 (1.80) | -32.1 (2.48)
Statistical Analysis 1: Comparison: ABT-335 + 10 mg Rosuvastatin vs 10 mg Rosuvastatin; An n = 205 per arm would provide >99% power to detect a 17% decrease in triglycerides relative to statin monotherapy for each combo therapy dose, assuming an SD of 30%; Test type: Superiority or Other; p < 0.001, ANCOVA — alpha = 0.05, all 3 primary endpoints had to show superiority of combo therapy in order to declare combo therapy successful at a given statin dose, Hochberg method for multiple comparison adjustment for 2 statin doses
Statistical Analysis 2: Comparison: ABT-335 + 20 mg Rosuvastatin vs 20 mg Rosuvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Final Visit
Description: [(Week 12 HDL-C minus baseline HDL-C)/baseline HDL-C] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline HDL-C value and at least 1 postbaseline HDL-C value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 224 | 225 | 220 | 239 | 236 | 115
percent change | 20.3 (1.36) | 19.0 (1.35) | 15.0 (1.37) | 8.5 (1.32) | 10.3 (1.32) | 9.3 (1.85)
Statistical Analysis 1: Comparison: ABT-335 + 10 mg Rosuvastatin vs 10 mg Rosuvastatin; An n = 205 per arm would provide 92% power to detect a 5% increase in HDL-C relative to statin monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 20 mg Rosuvastatin vs 20 mg Rosuvastatin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Final Visit
Description: [(Week 12 LDL-C minus baseline LDL-C)/baseline LDL-C] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline LDL-C value and at least 1 postbaseline LDL-C value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 231 | 230 | 223 | 243 | 238 | 120
percent change | -37.2 (1.21) | -38.8 (1.21) | -6.5 (1.22) | -38.0 (1.18) | -45.0 (1.19) | -50.6 (1.64)
Statistical Analysis 1: Comparison: ABT-335 + 10 mg Rosuvastatin vs ABT-335; An n = 205 per arm would provide 99% power to detect a 43% decrease in LDL-C relative to ABT-335 monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 20 mg Rosuvastatin vs ABT-335; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Percent Change in Non-low-density Lipoprotein Cholesterol (Non-HDL-C)From Baseline to Final Visit
Description: [(Week 12 non-HDL-C minus baseline non-HDL-C)/baseline non-HDL-C] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline non-HDL-C value and at least 1 postbaseline non-HDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 224 | 225 | 220 | 238 | 236 | 115
percent change | -44.7 (1.05) | -45.3 (1.04) | -18.5 (1.06) | -39.8 (1.02) | -45.8 (1.02) | -51.5 (1.43)

5. Secondary Outcome: Mean Percent Change in Very Low-density Lipoprotein Cholesterol (VLDL-C) From Baseline to Final Visit
Description: [(Week 12 VLDL-C minus baseline VLDL-C)/baseline VLDL-C] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline VLDL-C value and at least 1 postbaseline VLDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 243 | 237 | 235 | 244 | 243 | 126
percent change | -55.8 (3.08) | -50.6 (3.10) | -31.9 (3.13) | -41.0 (3.07) | -42.1 (3.07) | -49.1 (4.17)

6. Secondary Outcome: Mean Percent Change in Total Cholesterol From Baseline to Final Visit
Description: [(Week 12 total cholesterol minus baseline total cholesterol)/baseline total cholesterol] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline total cholesterol value and at least 1 postbaseline total cholesterol value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 252 | 249 | 242 | 252 | 255 | 127
percent change | -34.4 (0.82) | -35.7 (0.83) | -13.5 (0.84) | -32.5 (0.82) | -37.3 (0.82) | -42.7 (1.13)

7. Secondary Outcome: Mean Percent Change in Lipoprotein Apo B (Apo B) From Baseline to Final Visit
Description: [(Week 12 Apo B minus baseline Apo B)/baseline Apo B] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline ApoB and at least 1 postbaseline ApoB value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 252 | 244 | 239 | 248 | 252 | 123
percent change | -39.2 (1.04) | -39.2 (1.05) | -16.2 (1.06) | -34.1 (1.04) | -39.6 (1.03) | -45.0 (1.45)

8. Secondary Outcome: Median Percent Change in High-sensitivity C-reactive Protein (hsCRP) From Baseline to Final Visit
Description: [(Week 12 hsCRP minus baseline hsCRP)/baseline hsCRP] x 100
Time Frame: Baseline to 12 Weeks
Population: All randomized subjects with a baseline hsCRP value and at least 1 postbaseline hsCRP value, LOCF
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Number analyzed (Participants) | 252 | 246 | 241 | 249 | 254 | 125
percent change | -33.8 (16.87) [-52.4 to 0.2] | -40.8 (17.01) [-59.9 to -10.3] | -12.1 (17.20) [-40.1 to 22.7] | -22.9 (16.92) [-48.1 to 12.3] | -29.9 (16.78) [-53.8 to 4.1] | -33.1 (23.31) [-59.0 to -6.4]

ADVERSE EVENTS:
Arm/Group | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 10 | 3 | 10 | 3 | 7 | 2
Other Adverse Events (participants affected / at risk) | 126 | 114 | 117 | 109 | 110 | 61
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Coronary artery disease (Cardiac disorders) | 1/261 | 1/261 | 1/259 | 0/261 | 1/266 | 0/131
Myocardial infarction (Cardiac disorders) | 2/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Myocardial ischaemia (Cardiac disorders) | 0/261 | 1/261 | 0/259 | 0/261 | 0/266 | 0/131
Pericarditis (Cardiac disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Colitis (Gastrointestinal disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0/261 | 0/261 | 0/259 | 1/261 | 0/266 | 0/131
Pancreatitis acute (Gastrointestinal disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Chest pain (General disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Non-cardiac chest pain (General disorders) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Bronchitis (Infections and infestations) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Diverticulitis (Gastrointestinal disorders) | 0/261 | 1/261 | 1/259 | 0/261 | 0/266 | 0/131
Gastroenteritis (Infections and infestations) | 1/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Kidney infection (Infections and infestations) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Pneumonia (Infections and infestations) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Pyothorax (Infections and infestations) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Sepsis (Infections and infestations) | 0/261 | 0/261 | 0/259 | 1/261 | 0/266 | 0/131
Septic shock (Infections and infestations) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Urinary tract infection (Infections and infestations) | 0/261 | 0/261 | 0/259 | 1/261 | 0/266 | 0/131
Back pain (Musculoskeletal and connective tissue disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/261 | 0/261 | 2/259 | 0/261 | 0/266 | 0/131
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Guillain-Barre syndrome (Nervous system disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Presyncope (Nervous system disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Syncope (Nervous system disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Nephrolithiasis (Renal and urinary disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 1/266 | 0/131
Renal failure (Renal and urinary disorders) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Renal pain (Renal and urinary disorders) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 0/131
Vaginal prolapse (Reproductive system and breast disorders) | 0/261 | 0/261 | 0/259 | 0/261 | 0/266 | 1/131
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/261 | 0/261 | 0/259 | 1/261 | 0/266 | 0/131
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/261 | 0/261 | 0/259 | 0/261 | 0/266 | 0/131
Peripheral vascular disorder (Vascular disorders) | 0/261 | 0/261 | 1/259 | 0/261 | 0/266 | 1/131
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | ABT-335 + 10 mg Rosuvastatin | ABT-335 + 20 mg Rosuvastatin | ABT-335 | 10 mg Rosuvastatin | 20 mg Rosuvastatin | 40 mg Rosuvastatin
Constipation (Gastrointestinal disorders) | 11/261 | 7/261 | 9/259 | 6/261 | 9/266 | 4/131
Diarrhea (Gastrointestinal disorders) | 7/261 | 8/261 | 7/259 | 6/261 | 8/266 | 6/131
Dyspepsia (Gastrointestinal disorders) | 5/261 | 13/261 | 9/259 | 9/261 | 7/266 | 5/131
Nausea (Gastrointestinal disorders) | 9/261 | 14/261 | 12/259 | 12/261 | 11/266 | 5/131
Stomach discomfort (Gastrointestinal disorders) | 3/261 | 2/261 | 3/259 | 5/261 | 3/266 | 5/131
Fatigue (General disorders) | 12/261 | 12/261 | 6/259 | 7/261 | 7/266 | 4/131
Pain (General disorders) | 7/261 | 2/261 | 8/259 | 7/261 | 2/266 | 6/131
Nasopharyngitis (Infections and infestations) | 10/261 | 9/261 | 6/259 | 14/261 | 8/266 | 5/131
Sinusitis (Infections and infestations) | 9/261 | 6/261 | 10/259 | 2/261 | 3/266 | 3/131
Upper respiratiory tract infection (Infections and infestations) | 12/261 | 12/261 | 10/259 | 5/261 | 6/266 | 4/131
Alanine aminotransferase increased (Investigations) | 4/261 | 9/261 | 4/259 | 2/261 | 2/266 | 2/131
Aspartate aminotransferase increased (Investigations) | 4/261 | 8/261 | 3/259 | 2/261 | 1/266 | 2/131
Blood creatine phosphokinase increased (Investigations) | 5/261 | 5/261 | 4/259 | 3/261 | 7/266 | 4/131
Arthralgia (Musculoskeletal and connective tissue disorders) | 11/261 | 8/261 | 10/259 | 10/261 | 9/266 | 9/131
Back pain (Musculoskeletal and connective tissue disorders) | 15/261 | 15/261 | 17/259 | 17/261 | 16/266 | 6/131
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7/261 | 6/261 | 3/259 | 10/261 | 12/266 | 4/131
Myalgia (Musculoskeletal and connective tissue disorders) | 10/261 | 7/261 | 7/259 | 15/261 | 9/266 | 9/131
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/261 | 2/261 | 3/259 | 1/261 | 0/266 | 4/131
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5/261 | 8/261 | 14/259 | 14/261 | 9/266 | 6/131
Dizziness (Nervous system disorders) | 12/261 | 9/261 | 12/259 | 4/261 | 6/266 | 0/131
Headache (Nervous system disorders) | 40/261 | 23/261 | 30/259 | 33/261 | 44/266 | 20/131
Insomnia (Psychiatric disorders) | 6/261 | 8/261 | 6/259 | 3/261 | 3/266 | 3/131
Cough (Respiratory, thoracic and mediastinal disorders) | 6/261 | 4/261 | 6/259 | 3/261 | 1/266 | 4/131
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3/261 | 2/261 | 3/259 | 7/261 | 3/266 | 4/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall be so restricted after the expiration of twelve (12) months from completion of the studies at all sites. Any presentation or publication to be submitted to Sponsor (in draft of the same) for Sponsor review and comment.